CLINICAL TRIAL: NCT05497401
Title: A Controlled Study to Evaluate the Efficacy of Allogeneic MesenCure for the Treatment of Patients With ARDS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BonusBio Group Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCS-03
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-12

CONDITIONS: ARDS

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment (Experimental)
  Interventions: Biological: MesenCure
- control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MesenCure — Enhanced mesenchymal cell-based product
  Arms: treatment
Other: Placebo — Saline
  Arms: control

SUMMARY:
The efficacy of the allogeneic cell-therapy product MesenCure in addition to standard of care will be evaluated in comparison to placebo control in 300 moderate to severe Covid patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients are able and agree to sign informed consent form before any study-specific procedure.
2. Males or females, age range 18-80.
3. Documented ARDS
4. RA-O2 Saturation of ≤93% and/or Evidence of COVID19-related pulmonary infiltrates on chest X-ray/thoracic tomography
5. Stable hemodynamic condition (blood pressure of systolic <180mm Hg and diastolic <110mm Hg)

Exclusion Criteria:

General:

1. Pregnant or breast-feeding females.
2. History of drug abuse.
3. Heavy smokers (above 2 packages a day).
4. Subjects incapable of giving consent.

Background medical conditions:

1. Known history of any significant medical disorder, which in the investigator's judgment contraindicates the subject's participation.
2. History of advanced congestive heart failure or active acute myocardial infarction (AMI), renal failure (estimated GFR of <30 ml/min/1.73 m2 at screening), or hepatic disease (hepatic insufficiency classified as Child-Pugh B or C).
3. Known autoimmune diseases.
4. Received any investigational drug within 30 days prior to screening day (Visit 1) (Remdesivir is not considered investigational, and is not an exclusion criteria).
5. Immunocompromised condition from any reason, at screening.
6. Abnormal clinically significant laboratory test findings, as per the investigator's judgment.
7. Poorly controlled diabetic subjects (HbA1c > 9%).
8. Known active lung malignancy.

Concomitant treatment:

1. Currently treated with Immunosuppressive agents other than corticosteroids used for treating COVID19.
2. Treatment for cancer (i.e. chemotherapy or radiotherapy treatment) within the last 12 months.

Hypersensitivity:

1. Known history of hypersensitivity to Dextran-40.
2. Known history of hypersensitivity to Human Serum Albumin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 month
CRP reduction | 14 days
  Blood CRP is measured in mg/dL
Invasive ventilation | 1 month

IPD SHARING:
Plan to Share IPD: No